CLINICAL TRIAL: NCT03015948
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Dose of SHR4640 in Healthy Male Volunteers
Brief Title: A Single Dose Study of SHR4640 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SHR4640-101-AUS
Record Dates: First submitted 2016-09-20; First posted 2017-01-10 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — ruzinurad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 2.5mg SHR4640 (Experimental): 10 subjects will be randomized in a 4:1 ratio to receive a single dose of either 2.5 mg SHR4640 (n=8) or placebo (n=2)
  Interventions: Drug: SHR4640
- 10mg SHR4640 (Experimental): 10 subjects will be randomized in a 4:1 ratio to receive a single dose of either 10mg SHR4640 (n=8) or placebo (n=2) 10mg.
  Interventions: Drug: SHR4640
- 20mg SHR4640 (Experimental): 10 subjects will be randomized in a 4:1 ratio to receive a single dose of either 20mg SHR4640 (n=8) or placebo (n=2) .
  Interventions: Drug: SHR4640
- Placebo (Experimental): For each dose cohort, 10 subjects will be randomized in a 4:1 ratio to receive a single dose of either SHR4640 (n=8) or placebo (n=2)
  Interventions: Drug: Placebo
- 5mg SHR4640 (Experimental): 10 subjects will be randomized in a 4:1 ratio to receive a single dose of either 5 mg SHR4640 (n=8) or placebo (n=2)
  Interventions: Drug: SHR4640

INTERVENTIONS:
Drug: SHR4640 — a single dose of SHR4640 (n=8) for each dose cohort
  Arms: 10mg SHR4640; 2.5mg SHR4640; 20mg SHR4640; 5mg SHR4640
Drug: Placebo — a single dose of placebo (n=2) for each dose cohort .
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, single ascending-dose Phase I trial.

DETAILED DESCRIPTION:
This study includes screening (Days -16 to -3), check-in (Day -2), enrollment (Day -1), dosing (Day 1), observational period (Days 2 to 3), discharge day (Day 4), and safety follow-up visit (Day 8). Forty eligible subjects will be enrolled into 4 dose cohorts (10 for each cohort), and every 10 subjects will be randomized in a 4:1 ratio to receive a single dose of either SHR4640 (n=8) or placebo (n=2).

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged between 18 and 55 years, inclusive.
2. Body weight ≥ 50 kg and body mass index between 18.0 to 30.0 kg/m2, inclusive.
3. Screening sUA level from 0.24 to 0.42 mmol/L, inclusive.
4. Considered generally healthy upon completion of medical history, full physical examination, vital signs, laboratory parameters (including thyroid function, coagulation and serological tests, hematology, creatinine kinase, biochemistry, and urinalysis), 12-lead ECG, and abdominal ultrasound, as judged by the Investigator.
5. Agrees to use a highly effective method of contraception, i.e. condom and suitable contraception for your female partner e.g. diaphragm (double barrier), oral contraceptive or intrauterine contraceptive device during heterosexual intercourse or be non-heterosexually active, or practice sexual abstinence throughout the study period and for 30 days following study drug dosing, and must agree to refrain from sperm donation from Day -2 until at least 30 days following study drug dosing.
6. Negative drug screen (including alcohol) at screening and on admission to clinical site.
7. Able to understand the study procedures and the risks involved and must be willing to provide written informed consent before any study-related activity.

Exclusion Criteria:

1. History of hypersensitivity to SHR4640 or its analogues.
2. Screening sCr above upper limit of normal.
3. Screening alanine aminotransferase, aspartate aminotransferase, total bilirubin, or gamma glutamyl transferase > 1.5 × upper limit of normal.
4. Positive result for HIV.
5. Positive result for hepatitis B surface antigen or hepatitis C virus antibody.
6. History or presence of kidney stones.
7. Acute or chronic illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial product to the subject.
8. Undergone major surgery within 3 months of Day 1.
9. Donated any blood or plasma in the past month or more than 400 mL within 3 months of Day 1.
10. Has poor venous access and is unable to donate blood.
11. Use of tobacco products within 30 days of Day 1.
12. Heavy caffeine drinker (more than 5 cups or glasses of caffeinated beverages per day).
13. History of drug and/or alcohol abuse in the last year.
14. Consumes more than 14 drinks of alcohol per week (eg, 1 drink = 5 oz [150 mL] of wine, 12 oz of beer, or 1.5 oz of hard liquor).
15. Consumes grapefruit and/or poppy seed within 5 days of Day 1.
16. Cannot refrain from heavy exercises, tobacco products, alcohol, grapefruit, and/or poppy seed from Day -2 to Day 4.
17. Use of any of the following, unless agreed as nonclinically relevant by the Investigator and the Sponsor:

1) Prescription medication within 2 weeks of Day 1. 2) Over-the-counter medication within 1 week of Day 1. 3) Use of any over the-counter, nutraceuticals, or prescription medications that might interfere with the absorption, distribution, metabolism, or excretion of SHR4640 (proton-pump inhibitor, fluconazole, indomethacin, ranitidine, flurbiprofen, probenecid, aprepitant, etc.) within 1 month of Day 1.

18. Received the last dose of a study drug (or treatment with a medical device) within 30 days or 5 T1/2 (whichever is longer) of the study drug of Day 1 or are currently participating in another study of a study drug (or medical device).

19. Any other medical or psychological condition, which in the opinion of the Investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements or to complete the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2016-11-23 (Actual)

PRIMARY OUTCOMES:
Assess safety and tolerability of SHR 4640 over 11days including AEs, laboratory safety variables (including hematology, creatinine kinase (CK), biochemistry, and urinalysis), physical examinations, vital signs, and 12-lead electrocardiograms (ECGs) | 11 days

SECONDARY OUTCOMES:
Assess Pharmacokinetics (PK) Plasma parameter Area under the concentration-time curve (AUC) from zero to 24 and 72 hours postdose and from zero to infinity. | from time of dosing to 72 hours
Assess Pharmacokinetics (PK) Plasma parameter Time to maximum concentration. | from time of dosing to 72 hours
Assess Pharmacokinetics (PK) Plasma parameter Maximum concentration. | from time of dosing to 72 hours
Assess Pharmacokinetics (PK) Plasma parameter Terminal elimination half-life (T1/2). | from time of dosing to 72 hours
Assess Pharmacodynamics (PD) parameter Actual and percent changes in serum uric acid (sUA )from baseline. | from time of dosing to 72 hours
Assess Pharmacodynamics (PD) parameter urinary uric acid concentration (uUA): actual and percent changes from baseline. | from time of dosing to 72 hours
Assess Pharmacodynamics (PD) parameter urinary uric acid excretion (eUA): actual and percent changes from baseline. | from time of dosing to 72 hours
Assess Pharmacodynamics (PD) parameter Uric acid renal clearance (UaCl): actual and percent changes from baseline | from time of dosing to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sam Salman, B.Sc,BMBS, Principal Investigator — Linear Clinical Research
Locations (1):
- Atridia Pty Limited, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No